CLINICAL TRIAL: NCT00248716
Title: Treatment of Anemia in the 2nd Year of Life. Comparison of the Efficacy of Two Different Iron Preparations.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Dr Jacob Urkin, Ben-Gurion University of the Negev
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sor458607ctil
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2008-04

CONDITIONS: Iron Deficiency; Anemia
MeSH Terms: conditions — Iron Deficiencies; Anemia | interventions — ferrous gluconate; Niferex

INTERVENTIONS:
Drug: Ferrous gluconate and iron polysaccharide complex — Children with anemia will receive 5mg per kg per day of one of study medications. Treatment period for 3 months

SUMMARY:
Healthy toddlers (age 9-18 month) following a routine blood count will be placed in three groups:

1. Iron deficiency with no anemia
2. anemia
3. no anemia and no iron deficiency Following a nutritional questionnaire, parents of all toddlers will receive instruction regarding appropriate nutrition in the 2nd year of life. Groups 1 and 2 will randomly receive one of two preparations currently in use for treatment of iron deficiency in Israel (Aktiron 35 - Ferrous gluconate and Ferripel-3 - iron polysaccharide complex). Followup blood count will be taken 3 month after recruitment. The study aims to compare the effectiveness of the Iron preparations regarding compliance and efficacy.

The hypothesis is that a significant difference will be detected between the two preparations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy toddlers age 9-18 months

Exclusion Criteria:

* Toddlers with: chronic diseases, prematurity, inherited hematological disease.

Ages: 9 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Urkin, MD, MPH, Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Primary Pediatric Care Unit, Ben-Gurion University of the Negev, Beersheba, Israel